CLINICAL TRIAL: NCT04775810
Title: Pilot Study of a Signal-processing Algorithm Aiming at Improving Speech-in-noise Intelligibility in Normal-hearing and Hearing-impaired Persons
Brief Title: Study of a Signal-processing Algorithm Aiming at Improving Speech-in-noise Intelligibility in Normal-hearing and Hearing-impaired Persons
Acronym: AUDIOCAP 1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Archean Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUDIOCAP_CT01; 2020-A02253-36 (Other: ID-RCB)
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Speech Intelligibility in Noise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The device is an algorithm designed to enhance speech intelligibility of speech-in-noise signals — Normal-hearing and hearing-impaired subjects will listen to speech-in-noise audio files that are either unprocessed or processed in order to increase speech intelligibility.

SUMMARY:
Nearly half a billion people suffer from disabling hearing loss. The most common form of hearing loss in adults is age-related hearing loss (ARHL), which causes a reduced ability to understand speech in noisy environments. The ability of people with ARHL to communicate is therefore greatly impacted, limiting their social interactions and thus their quality of life. Yet, the wear of hearing aids - which is the current standard rehabilitation treatment in such cases - does not lead to optimal satisfactory outcomes when it comes to understanding speech in noisy environments.

The objective of this pilot study is to test a new signal-processing algorithm, based on artificial intelligence, that aims at enhancing the intelligibility of speech-in-noise signals. The efficiency of the algorithm is compared to a standard denoising algorithm commonly used in hearing aids. The primary outcome measure is the word-identification performance of the participants, using the FrMatrix test (Jansen et al., 2012). Two secondary outcome measures are investigated: listening effort (self-assessed using a Likert scale, and measured through response times), and subjective preference (assessed in a paired-comparison task).

The study is conducted in 20 normal-hearing subjects and in 40 older (age ≥ 55 years) hearing-impaired subjects.

ELIGIBILITY:
Inclusion criteria for normal-hearing participants :

* consenting to and available for the study
* age ≥ 18 years and ≤ 25 years
* right-handed
* native French speaker
* pure-tone air-conduction audiometric thresholds at .5, 1, 2, and 4 kHz all ≤ 20 dB hearing loss (HL)

Exclusion criteria for normal-hearing participants :

* score at the Tinnitus Handicap Inventory > 56
* uncorrected visual impairment
* pregnancy
* subject placed under legal authority (guardianship, tutorship)

Inclusion criteria for hearing-impaired participants :

* consenting to and available for the study
* age ≥ 55 years
* native French speaker
* pure-tone air-conduction average hearing thresholds (PTA) for frequencies of .5, 1, 2, and 4 kHz ≥ 30 dB HL and ≤ 70 dB HL
* right-ear PTA for low frequencies (< 2 kHz) lower than the right-ear PTA for high frequencies (> 4 kHz). The difference between the two PTAs must be ≥ 20 dB
* the difference between the PTA for frequencies of .5, 1, 2, and 4 kHz (PTA.5-4kHz) in the right ear and the left-ear PTA.5-4kHz must be ≤ 10 dB

Exclusion criteria for hearing-impaired participants :

* score at the Tinnitus Handicap Inventory > 56
* history of a hearing impairment that was left uncorrected for more than 10 years
* uncorrected visual impairment
* congenital hearing impairment
* Ménière's disease
* auditory neuropathy
* mixed hearing loss
* fluctuating hearing impairment
* sudden hearing loss
* hearing impairment concomitant with other symptoms (e.g. vertigo)
* score at the Montreal Cognitive Assessment (MoCA) < 27
* subject placed under legal authority (guardianship, tutorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Speech-in-noise word identification | during procedure, T1
  Speech-in-noise word identification score as assessed using the FrMatrix test

SECONDARY OUTCOMES:
Listening effort | during procedure, T1
  response times recorded during the FrMatrix test
Listening effort | during procedure, T1
  self-assessed subjective measures of listening effort.
Subjective preference in terms of speech naturalness | during procedure, T1
  Measures of relative preference using forced-choice pairwise comparisons

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Rive Gauche, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amieva H, Ouvrard C, Giulioli C, Meillon C, Rullier L, Dartigues JF. Self-Reported Hearing Loss, Hearing Aids, and Cognitive Decline in Elderly Adults: A 25-Year Study. J Am Geriatr Soc. 2015 Oct;63(10):2099-104. doi: 10.1111/jgs.13649. PMID 26480972
- [Background] Bentler RA. Effectiveness of directional microphones and noise reduction schemes in hearing aids: a systematic review of the evidence. J Am Acad Audiol. 2005 Jul-Aug;16(7):473-84. doi: 10.3766/jaaa.16.7.7. PMID 16295234
- [Background] Chong FY, Jenstad LM. A critical review of hearing-aid single-microphone noise-reduction studies in adults and children. Disabil Rehabil Assist Technol. 2018 Aug;13(6):600-608. doi: 10.1080/17483107.2017.1392619. Epub 2017 Oct 26. PMID 29072542
- [Background] Ciorba A, Bianchini C, Pelucchi S, Pastore A. The impact of hearing loss on the quality of life of elderly adults. Clin Interv Aging. 2012;7:159-63. doi: 10.2147/CIA.S26059. Epub 2012 Jun 15. PMID 22791988
- [Background] Ghulyan-Bedikian V, Paolino M, Giorgetti-D'Esclercs F, Paolino F. [Psychometric properties of a French adaptation of the Tinnitus Handicap Inventory]. Encephale. 2010 Oct;36(5):390-6. doi: 10.1016/j.encep.2009.12.007. Epub 2010 Jan 27. French. PMID 21035629
- [Background] Gonthier C, Thomassin N, Roulin JL. The composite complex span: French validation of a short working memory task. Behav Res Methods. 2016 Mar;48(1):233-42. doi: 10.3758/s13428-015-0566-3. PMID 25669761
- [Background] Jansen S, Luts H, Wagener KC, Kollmeier B, Del Rio M, Dauman R, James C, Fraysse B, Vormes E, Frachet B, Wouters J, van Wieringen A. Comparison of three types of French speech-in-noise tests: a multi-center study. Int J Audiol. 2012 Mar;51(3):164-73. doi: 10.3109/14992027.2011.633568. Epub 2011 Nov 28. PMID 22122354
- [Background] Krueger M, Schulte M, Zokoll MA, Wagener KC, Meis M, Brand T, Holube I. Relation Between Listening Effort and Speech Intelligibility in Noise. Am J Audiol. 2017 Oct 12;26(3S):378-392. doi: 10.1044/2017_AJA-16-0136. PMID 29049622
- [Background] Lakshmi MSK, Rout A, O'Donoghue CR. A systematic review and meta-analysis of digital noise reduction hearing aids in adults. Disabil Rehabil Assist Technol. 2021 Feb;16(2):120-129. doi: 10.1080/17483107.2019.1642394. Epub 2019 Sep 10. PMID 31502900
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Mener DJ, Betz J, Genther DJ, Chen D, Lin FR. Hearing loss and depression in older adults. J Am Geriatr Soc. 2013 Sep;61(9):1627-9. doi: 10.1111/jgs.12429. No abstract available. PMID 24028365
- [Background] Mick P, Kawachi I, Lin FR. The association between hearing loss and social isolation in older adults. Otolaryngol Head Neck Surg. 2014 Mar;150(3):378-84. doi: 10.1177/0194599813518021. Epub 2014 Jan 2. PMID 24384545
- [Background] Moore BC, Fullgrabe C, Stone MA. Determination of preferred parameters for multichannel compression using individually fitted simulated hearing AIDS and paired comparisons. Ear Hear. 2011 Sep-Oct;32(5):556-68. doi: 10.1097/AUD.0b013e31820b5f4c. PMID 21285878
- [Background] Moulin A, Richard C. Sources of variability of speech, spatial, and qualities of hearing scale (SSQ) scores in normal-hearing and hearing-impaired populations. Int J Audiol. 2016;55(2):101-9. doi: 10.3109/14992027.2015.1104734. Epub 2015 Dec 1. PMID 26624277
- [Background] Nasreddine ZS, Patel BB. Validation of Montreal Cognitive Assessment, MoCA, Alternate French Versions. Can J Neurol Sci. 2016 Sep;43(5):665-71. doi: 10.1017/cjn.2016.273. PMID 27670209
- [Background] Neher T, Grimm G, Hohmann V, Kollmeier B. Do hearing loss and cognitive function modulate benefit from different binaural noise-reduction settings? Ear Hear. 2014 May-Jun;35(3):e52-62. doi: 10.1097/AUD.0000000000000003. PMID 24351610
- [Background] Oldfield RC. The assessment and analysis of handedness: the Edinburgh inventory. Neuropsychologia. 1971 Mar;9(1):97-113. doi: 10.1016/0028-3932(71)90067-4. No abstract available. PMID 5146491
- See also: Anovum (2018). EuroTrak 2018. (Rapport). — https://www.ehima.com/wp-content/uploads/2018/07/EuroTrak_2018_FRANCE.pdf
- See also: WHO (2017). Global costs of unaddressed hearing loss and cost-effectiveness of interventions — https://apps.who.int/iris/bitstream/handle/10665/254659/9789241512046-eng.pdf
- See also: WHO (2020). Deafness and Hearing Loss. (Rapport) — https://www.who.int/news-room/fact-sheets/detail/deafness-and-hearing-loss